CLINICAL TRIAL: NCT04048707
Title: Angiotensin 2 as a Novel Treatment for Hepatorenal Syndrome
Brief Title: Angiotensin 2 for Hepatorenal Syndrome
Acronym: ANTHEM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding issues; the study was never started
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #19-005718
Record Dates: First submitted 2019-07-29; First posted 2019-08-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Hepatorenal Syndrome; Cirrhosis; Kidney Failure, Acute
MeSH Terms: conditions — Hepatorenal Syndrome; Fibrosis; Acute Kidney Injury | interventions — Angiotensin II; Giapreza; Midodrine; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Midodrine/Octreotide (Active Comparator): This arm will receive standard of care treatment of midodrine, octreotide, and albumin.
  Interventions: Drug: Midodrine; Drug: Octreotide; Drug: Albumin solution
- Angiotensin 2 (Experimental): This arm will receive the experimental treatment of angiotensin 2 infusion and albumin.
  Interventions: Drug: Angiotensin II; Drug: Albumin solution

INTERVENTIONS:
Drug: Angiotensin II — Intravenous
  Other Names: Giapreza
  Arms: Angiotensin 2
Drug: Midodrine — Pill
  Arms: Midodrine/Octreotide
Drug: Octreotide — Subcutaneous
  Arms: Midodrine/Octreotide
Drug: Albumin solution — Intravenous suspension

SUMMARY:
Hepatorenal syndrome (HRS) is a disease in which patients with cirrhosis (end stage liver failure) develop secondary kidney injury and failure. The current treatment available in the United States is a combination of octreotide and midodrine, which are meant to decrease the release of those hormones and raise the blood pressure, respectively, which would increase blood flow to the kidneys. Angiotensin 2 (Ang2) is a new vasopressor drug that was approved by the FDA in December 2017 for patients with low blood pressure and has been shown to have similar effects to octreotide and midodrine.

This study will investigate whether Ang2 reverses HRS among patients admitted to the intensive care unit (ICU) at Ronald Reagan Medical Center. Our study population will be patients with HRS who are already or will be admitted to the ICU. HRS will be defined by new internationally accepted guidelines published by the International Club of Ascites. All patients who are consented will undergo an Ang2 response trial, where low-dose Ang2 will be administered for 4 hours to see how the patients respond. This will help us characterize the nature of the patients' kidney failure for later analysis. Patients will then be randomized into the control group or the study group. Patients in the control group will receive octreotide (a subcutaneous injection) and midodrine (an oral drug). Patients in the study group will continue receiving intravenous infusion of Ang2. Patients in both groups will also receive albumin, a protein found commonly in human blood. Treatment will continue in both groups for four days, until complete reversal of HRS, dialysis, or death.

Our primary outcome will be rate of reversal of HRS, defined as improvement in kidney function.

ELIGIBILITY:
Inclusion Criteria: Patients in the ICU with HRS-AKI defined as

* Acute kidney injury defined as an increase in serum creatinine (sCr) >=0.3 mg/dl or >=50% from baseline within 7 days
* Presence of cirrhosis and ascites
* Absence of other causes such as shock, nephrotoxic drugs, or other suspected causes of kidney injury.
* Lack of response to diuretic withdrawal and albumin challenge of 1 g/kg of body weight

Exclusion Criteria:

* Age <18 years
* Current or anticipated (within 24 hours) need for renal replacement therapy (RRT)
* Cr > 6 mg/dl
* Renal transplantation status
* Fractional Excretion of Sodium (FeNa) > 2%
* Pregnancy
* Recent Cerebrovascular Accident (CVA), Myocardial Infarction (MI), venous or arterial thrombosis (within last 3 months)
* Known hypercoagulable state other than cirrhosis
* Uncontrolled hypertension (SBP > 160)
* Anticipated mortality within 72 hours
* Inability to obtain consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Reversal of hepatorenal syndrome | 4 days
  Partial or complete reversal of HRS. Serum creatinine will be measured daily and compared against the patient's baseline creatinine.
  Partial reversal is defined defined as improvement of at least one AKI stage as defined by International Club of Ascites Acute Kidney Injury (ICA-AKI) criteria Complete defined as improvement of serum creatinine to within 0.3 mg/dl of baseline value).
  ICA-AKI criteria:
  * Stage 1: increase in sCr ≥0.3 mg/dl (26.5 μmol/L) or an increase in sCr ≥1.5-fold to 2-fold from baseline
  * Stage 2: increase in sCr >2-fold to 3-fold from baseline
  * Stage 3: increase of sCr >3-fold from baseline or sCr ≥4.0 mg/dl (353.6 μmol/L) with an acute increase ≥0.3 mg/dl (26.5 μmol/L) or initiation of renal replacement therapy Angeli P et al. J Hepatology 2015:62(968-974)

SECONDARY OUTCOMES:
Need for renal replacement therapy | 4 days
  The treating team with the assistance of nephrology will assess the acute need for dialysis on a daily basis. If the patient does require urgent hemodialysis at their determination, this will be noted. The proportion of each group who required hemodialysis will be compared.
Mortality | 28 days
  In-hospital mortality
Serum sodium | 4 days
  Change in serum sodium from the beginning of the study to the end of the study.
Relapse of hepatorenal syndrome | 14 days
  Recurrence of HRS-AKI after withdrawal of study drug, defined as a worsening of AKI by at least one stage according to ICA-AKI criteria AKI grade as defined by ICA-AKI criteria (J Hepatology 2015:62[968-974])

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tumlin JA, Murugan R, Deane AM, Ostermann M, Busse LW, Ham KR, Kashani K, Szerlip HM, Prowle JR, Bihorac A, Finkel KW, Zarbock A, Forni LG, Lynch SJ, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Bellomo R; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Outcomes in Patients with Vasodilatory Shock and Renal Replacement Therapy Treated with Intravenous Angiotensin II. Crit Care Med. 2018 Jun;46(6):949-957. doi: 10.1097/CCM.0000000000003092. PMID 29509568
- [Background] Khanna A, Ostermann M, Bellomo R. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Dec 28;377(26):2604. doi: 10.1056/NEJMc1714511. No abstract available. PMID 29281568